CLINICAL TRIAL: NCT02988557
Title: Evaluation of the Effect of an Inclined Plane on the Walking of Children With Cerebral Palsy: What Are the Paths for Rehabilitation?
Brief Title: Walking Inclined Plane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC16_0089
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Cerebral Palsy; Spastic Diplegia
Keywords: cerebral palsy; gait; slope; electromyography
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise Test

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treadmill (Experimental)
  Interventions: Procedure: walking on a treadmill with a sloped surface; Device: treadmill

INTERVENTIONS:
Procedure: walking on a treadmill with a sloped surface — walking on a treadmill with a sloped surface
Device: treadmill — walking on a treadmill with a sloped surface

SUMMARY:
The adaptations in kinematics and muscle activity, investigated by 3D gait analysis and dynamic electromyography recordings, will be studied in children with bilateral spastic cerebral palsy during level walking, and before and after a training on a treadmill with a sloped surface (7°). Data will be compared with those obtained in a sample of typically developing (TD) children (controls)

DETAILED DESCRIPTION:
15 CP children and 15 TD children aged 6 to 14 years will take part in this study. Dynamic EMG recordings will be performed as well as kinematic data assessments through a gait analysis system. Three different slopes will be assessed, using a treadmill. The primary outcome measure will be the minimal knee extension value in the stance phase. The changes in kinematics will be overall assessed through the Gait Profile Score (Baker et al.). The details in changes will be assessed through statistical parametric mapping (SPM). The changes in muscle activity induced by the slope will be investigated by statistical parametric mapping of the EMG or kinematic data.

ELIGIBILITY:
Inclusion Criteria for children with CP:

* age = 6-14 years old
* children with cerebral palsy: spastic type, bilateral involvement, forefoot initial contact and/or excessive knee flexion at mid-stance and/or decreased hip extension in late stance.
* GMFCS I or II,
* Score on Gillette scale between 8 and 10
* able to walk at least 10 min without help

Inclusion Criteria for TD children:

* age = 6-14 years old

Exclusion Criteria:

* botulinum toxin injection or lower limb surgery within the last year.
* Uncontrolled seizures

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
minimal knee extension in stance (kinematics) | 1 day (single evaluation)
  quantitative value of the extension (degree(s))

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France